CLINICAL TRIAL: NCT03654677
Title: A Randomized, Double-blind, Multi-center, Active Controlled, Parallel-designed, Phase III Clinical Trial to Evaluate the Immunogenicity and Safety of Inactivated Hepatitis A Vaccine in Healthy Youths Above 16 Years or Adults
Brief Title: To Evaluate the Immunogenicity and Safety of Inactivated Hepatitis A Vaccine (VITHA-A)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BR-HAV-CT-302
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2020-03

CONDITIONS: Hepatitis A Vaccine
Keywords: Hepatitis A Vaccine
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inactivated hepatitis A vaccine (Experimental): Inactivated hepatitis A virus antigen 500U(Name of viral strain: TZ84)
  Interventions: Biological: inactivated hepatitis A vaccine
- Havrix Inj (Active Comparator): 1440 ELISA/mL_Adult Inj.(Name of Viral strain: HM175 Inj)
  Interventions: Biological: Havrix Inj

INTERVENTIONS:
Biological: inactivated hepatitis A vaccine — A single dose of the test vaccine or the control vaccine in the form of pre-filled syringe is injected intramuscularly into the deltoid muscle (not to be injected into the gluteal region), and additional vaccination is performed using the same vaccine and the same method at 6 months after the first vaccination.
  Arms: inactivated hepatitis A vaccine
Biological: Havrix Inj — A single dose of the test vaccine or the control vaccine in the form of pre-filled syringe is injected intramuscularly into the deltoid muscle (not to be injected into the gluteal region), and additional vaccination is performed using the same vaccine and the same method at 6 months after the first vaccination.
  Arms: Havrix Inj

SUMMARY:
The objective of this study is to evaluate the safety and immunogenicity after one primary dose and one additional dose (administered twice at an interval of 6 months) of inactivated hepatitis A vaccine are administered in adolescents (16 years of age or older) or adults.

DETAILED DESCRIPTION:
For this, a two-group comparison study will be conducted using a previously approved inactivated hepatitis A vaccine (Havrix Inj., manufactured by GSK) as the control vaccine to prove that the immunogenicity of the test vaccine treatment group is not inferior to the control vaccine treatment group and to statistically confirm that there is no difference in safety.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 16 years or older on the day of the first vaccination
* No history of hepatitis A or having hepatitis A vaccination
* Provided consent to the participation in the study voluntarily after receiving explanations about the objective, method, effect, etc. of this clinical study
* Determined by the investigator to be able to be followed up during the study period

Exclusion Criteria:

* A positive result (Anti-HAV 20 IU/L or above) in an hepatitis A antibody test at the time of screening
* Positive hepatitis type B antigen at the time of screening
* The following blood test results at the time of screening

  * ALT: More than 1.5 times the upper limit of normal
  * AST: More than 1.5 times the upper limit of normal
  * Total bilirubin: More than 1.5 times the upper limit of normal
* Tympanic temperature of 38°C or above within 48 hours prior to the vaccination or on the day of vaccination
* Moderate to severe acute or chronic infectious disease on the day of vaccination
* History of sensitivity to the following drugs: neomycin, formaldehyde, gentamicin sulfate, any preventive vaccines
* Congenital or acquired immunodeficient disease, or receiving immunosuppressive therapy
* Received immunosuppressive dose of systemic corticosteroids therapy within 12weeks days before vaccination
* uncontrolled epilepsy or neurological disorders
* Administered with other vaccine within 4 weeks prior to the screening
* Planned with other vaccine within 4 weeks after the vaccination date
* Used immunoglobulin formulation or human plasma, or received a transfusion within 12 weeks prior to the screening
* Participated in another clinical study within 12 weeks prior to the screening, or currently participating
* Pregnant women or breast-feeding women
* Other reasons not specified above that, in the opinion of the principal investigator, may make the subject ineligible to participate in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | 1 month after the second vaccination
  Seroconversion criteria: Anti-HAV 20 IU/L or above

SECONDARY OUTCOMES:
Seroconversion rate | 1 month after the first vaccination
  Seroconversion rate at 1 month after the first vaccination

OTHER OUTCOMES:
Safety endpoint (Adverse events) | Approximately 12 months after a consent to the participation
  Adverse events observed within 30 minutes after vaccination, solicited adverse events/adverse drug reactions, and unsolicited adverse events/adverse drug reactions through a diary, serious adverse events/adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hyun Choi, Principal Investigator — Incheon St.Mary's Hospital
Locations (12):
- South Korea (12):
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul, Banpo-dong, Seocho-gu
  - The Catholic University of Korea, Incheon St.Mary's Hospital, Incheon, Bupyeong-gu
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si, Gyeonggi-do
  - The Catholic University of Korea,Uijeongbu St.Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - The Catholic University of Korea,Yeouido St.Mary's Hospital, Seoul, Yeongdeungpo-gu
  - Hallym University Medical Center, Seoul, Yeongdeungpo-gu
  - Soon chung hyang university hospita, Bucheon-si
  - Inje university Ilsan Paik hospital, Ilsan
  - Ewha Womans University Mokdong Hospital, Seoul
  - Hanyang university medical center, Seoul
  - Kyunghee university hospital, Seoul
  - Soon Chun Hyang university hospital, Seoul

IPD SHARING:
Plan to Share IPD: No